CLINICAL TRIAL: NCT00166647
Title: Evaluation of Thiopurine Methyltransferase Polymorphisms in the Hispanic Population
Brief Title: Thiopurine Methyltransferase Polymorphisms Evaluation
Status: Withdrawn | Type: Observational
Why Stopped: Observational Study should not be in CT.gov
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: PPRU-10728
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Cancer
Keywords: Cancer; Chemotherapy; Hematological disorder
MeSH Terms: conditions — Neoplasms; Hematologic Diseases | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood Sampling

SUMMARY:
The purpose of the study is to determine the frequency of allelic variants in TPMT in the Hispanic population and to compare the frequency in the Hispanic population with the Caucasian Population.

DETAILED DESCRIPTION:
Relatively few studies have been performed evaluating the variant allele frequencies in Spanish populations. To date, no studies evaluating the TPMT variant allele frequency in the Hispanic population have been reported. Hispanics are a growing part of the patient population treated in the United States. Characterization of the proportion of patients with variant genotypes in this population is important since Hispanic children represent a significant proportion of children being treated with thiopurines.

A single 3 cc heparinized blood sample will be obtained for TPMT genotyping. The sample will be obtained either simultaneously with a clinical sample, at the time of an otherwise medically indicated intravenous catheter placement or scavenged from excess blood remaining following clinical laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* All Hispanic children and adolescents diagnosed and treated at Texas Children's Cancer Center within the last 5 years for malignant diseases/cancer and non-malignant hematological disorders that necessitate chemotherapy
* All Hispanic children and adolescents who will be treated at Texas Children's Center for malignant diseases/cancer and non-malignant hematological disorders that will necessitate chemotherapy.

Exclusion Criteria:

* Any child or adolescent registering at Texas Children's Cancer Center and not requiring any form of therapy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Texas Children's Hospital, Houston, Texas, United States